CLINICAL TRIAL: NCT03280108
Title: Clinical Investigation of AcrySof® IQ PanOptix™ IOL Model TFNT00
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ILH297-C001
Record Dates: First submitted 2017-09-06; First posted 2017-09-12 (Actual); Results first posted 2019-10-10 (Actual); Last update posted 2019-10-10 (Actual); Status verified 2019-10

CONDITIONS: Cataract
Keywords: Intraocular lens; IOL
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Multifocal IOL (Experimental): AcrySof IQ PanOptix Multifocal IOL Model TFNT00 implanted in the capsular bag in the posterior chamber following cataract removal and intended for long-term use over the lifetime of the cataract patient. Both eyes will be implanted (bilateral implantation).
  Interventions: Device: AcrySof IQ PanOptix Multifocal IOL
- Monofocal IOL (Active Comparator): AcrySof Monofocal IOL Model SN60AT implanted in the capsular bag in the posterior chamber following cataract removal and intended for long-term use over the lifetime of the cataract patient. Both eyes will be implanted (bilateral implantation).
  Interventions: Device: AcrySof Monofocal IOL

INTERVENTIONS:
Device: AcrySof IQ PanOptix Multifocal IOL — AcrySof IQ PanOptix Multifocal IOL Model TFNT00 for near, intermediate, and distance vision
  Other Names: Model TFNT00; AcrySof® IQ PanOptix®
  Arms: Multifocal IOL
Device: AcrySof Monofocal IOL — AcrySof Monofocal IOL Model SN60AT for single vision
  Other Names: Model SN60AT; AcrySof®
  Arms: Monofocal IOL

SUMMARY:
The purpose of this clinical study is to compare the visual outcomes of the AcrySof IQ PanOptix Multifocal Intraocular Lens (IOL) Model TFNT00 against that of a monofocal lens, the AcrySof Monofocal IOL Model SN60AT, in order to demonstrate comparable distance vision and superior near and intermediate vision.

DETAILED DESCRIPTION:
Both eyes of a subject must require cataract surgery to qualify for enrollment into this study. Subjects participating in the trial will attend a total of 10 study visits over a 7-month period. Of these 10 visits, 1 is preoperative, 2 are operative, and the remaining 7 are postoperative visits. Primary endpoint data will be collected at the Month 6 (Day 120-180) post second eye implantation visit.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with bilateral cataracts with planned cataract removal by phacoemulsification with a clear cornea incision
* Able to comprehend and willing to sign informed consent and complete all required postoperative follow-up procedures
* Clear intraocular media other than cataract in both eyes.
* Preoperative keratometric astigmatism of less than 1.0 diopter (D) in both operative eyes.

Exclusion Criteria:

* Clinically significant corneal abnormalities including corneal dystrophy, irregularity, inflammation or edema
* Previous refractive surgery or refractive surgery procedures (including, but not limited to LASIK, astigmatic keratotomy, and limbal relaxing incisions)
* Glaucoma (uncontrolled or controlled with medication)
* Degenerative eye disorders (e.g. macular degeneration or other retinal disorders)
* Pregnant or lactating
* Expected to require a second surgical intervention or retinal laser treatment.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-09-27 (Actual); Study Completion 2018-09-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alcon Research, Study Director — Alcon Research
Locations (12):
- United States (12):
  - Alcon Investigative Site, Fresno, California
  - Alcon Investigative Site, Mt. Dora, Florida
  - Alcon Investigative Site, Panama City, Florida
  - Alcon Investigative Site, Poughkeepsie, New York
  - Alcon Investigative Site, Mt. Pleasant, South Carolina
  - Alcon Investigative Site, Sioux Falls, South Dakota
  - Alcon Investigative Site, Nashville, Tennessee
  - Alcon Investigative Site, Houston, Texas
  - Alcon Investigative Site, Hurst, Texas
  - Alcon Investigative Site, Nacogdoches, Texas
  - Alcon Investigative Site, Salt Lake City, Utah
  - Alcon Investigative Site, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 12 investigative sites located in the United States.
Pre-assignment Details: Of the 250 enrolled, 7 subjects were exited as screen failures prior to attempted implantation. This reporting group includes all subjects with at least one eye implanted (243).
Groups:
- TFNT00: AcrySof IQ PanOptix Multifocal IOL Model TFNT00 bilaterally implanted in the capsular bag in the posterior chamber following cataract removal.
- SN60AT: AcrySof Monofocal IOL Model SN60AT bilaterally implanted in the capsular bag in the posterior chamber following cataract removal.
Period: Overall Study
Arm/Group | TFNT00 | SN60AT
Started (Successful Implantation) | 129 | 114
Completed | 127 | 114
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 2 | 0

BASELINE CHARACTERISTICS:
Population: This analysis population includes all eyes with successful IOL implantation with at least 1 post-operative visit (All-Implanted Analysis Set).
Groups:
- Total: Total of all reporting groups
Arm/Group | TFNT00 | SN60AT | Total
Number analyzed (Participants) | 129 | 114 | 243
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.8 (7.31) | 69.0 (6.46) | 67.3 (7.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85 | 79 | 164
  Male | 44 | 35 | 79
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 113 | 96 | 209
  Black or African American | 8 | 11 | 19
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 7 | 1 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  Other | 1 | 4 | 5

OUTCOME MEASURES:

1. Primary Outcome: Mean Photopic Monocular Best Corrected Distance Visual Acuity (4 m)
Description: Visual acuity (VA) was tested monocularly (each eye separately) under photopic (well-lit) conditions using the correction obtained from the manifest refraction and 100% contrast electronic Early Treatment Diabetic Retinopathy Study (ETDRS) charts at a distance of 4 meters (m) from the eye. VA was measured in logarithm of the minimum angle of resolution (logMAR), with 0.02 logMAR increment corresponding to a single letter on an ETDRS chart. A lower numeric value represents better visual acuity. This analysis was prespecified for the first operative eye.
Time Frame: Month 6 (Day 120-180), post second eye implantation
Population: All-Implanted Analysis Set with data available at the visit
Measure: Least Squares Mean (Standard Error); unit: logMAR
Arm/Group | TFNT00 | SN60AT
Number analyzed (Participants) | 127 | 113
logMAR | -0.014 (0.0083) | -0.039 (0.0087)
Statistical Analysis 1: Comparison: TFNT00 vs SN60AT; Test type: Non-Inferiority — Non-inferiority based on the observed 95% Upper Confidence Limit of the difference in Least Squares Means (LSM) between the 2 groups (TFNT00 - SN60AT). Non-inferiority margin = 0.10 logMAR; Least Squares Mean Difference = 0.024, 95% CI 1-sided [upper limit 0.041], Standard Error of Mean 0.0103

2. Primary Outcome: Mean Photopic Monocular Distance Corrected Visual Acuity at Near (40 cm)
Description: VA was tested monocularly under photopic conditions using the manifest refraction adjusted for optical infinity and 100% contrast electronic ETDRS charts at a distance of 40 centimeters (cm) from the eye. Distance corrected visual acuity at near was measured in logMAR, with 0.02 logMAR increment corresponding to a single letter on an ETDRS chart. A lower numeric value represents better visual acuity. This analysis was prespecified for the first operative eye.
Time Frame: Month 6 (Day 120-180), post second eye implantation
Population: All-Implanted Analysis Set with data at visit
Measure: Least Squares Mean (Standard Error); unit: logMAR
Units Other Than Participants: Eyes
Arm/Group | TFNT00 | SN60AT
Number analyzed (Participants) | 127 | 113
Number analyzed (Eyes) | 127 | 113
logMAR | 0.105 (0.0119) | 0.529 (0.0127)
Statistical Analysis 1: Comparison: TFNT00 vs SN60AT; Test type: Superiority; p < 0.001, Mixed Models Analysis

3. Primary Outcome: Cumulative Rate of Secondary Surgical Interventions (SSI) Related to Optical Properties of the IOL, First Eye
Description: The number of SSI's related to the optical properties of the IOL was calculated from time of implantation up to Month 6. The percentage was calculated as (# of eyes with an SSI related to the optical properties of the IOL) divided by (# of eyes with attempted IOL implantation, successful or aborted after contact with the eye) times 100. SSI's could include, but were not limited to, IOL replacement, IOL explantation, IOL repositioning, refractive laser treatment, paracentesis, vitreous aspirations, iridectomy or laser iridotomy for pupillary block, wound leak repair, and retinal detachment repair. No hypothesis testing was planned for this outcome measure.
Time Frame: Up to Month 6 (Day 120-180), post second eye implantation
Population: This analysis population includes all eyes with attempted (successful or aborted after contact with the eye) IOL implantation (Safety Analysis Set).
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | TFNT00 | SN60AT
Number analyzed (Participants) | 129 | 114
Number analyzed (Eyes) | 129 | 114
Eyes | 1 | 0

4. Primary Outcome: Mean Photopic Without Glare Binocular Distance Contrast Sensitivity
Description: Contrast sensitivity (ie, the ability to detect objects by distinguishing them from their background) was assessed binocularly (both eyes together) with the subject's best spectacle correction under photopic (well-lit) conditions at a distance of 8 feet from the eye at spatial frequencies of 3, 6, and 12, and 18 cycles per degree (cpd) using the Vector Vision CSV 1000-HGT without a glare source. Raw scores from contrast sensitivity testing were transformed to log units. Subjects who were unable to see a targeted spatial frequency at any available contrast, including that of the reference patch, were assigned the lowest measurable value. A higher numeric value represents better contrast sensitivity. Hypothesis testing was not planned for this outcome measure.
Time Frame: Month 6 (Day 120-180), post second eye implantation
Population: Safety Analysis Set with contrast sensitivity test
Measure: Mean (Standard Deviation); unit: log units
Arm/Group | TFNT00 | SN60AT
Number analyzed (Participants) | 127 | 111
log units
  3 cpd | 1.752 (0.2080) | 1.733 (0.1989)
  6 cpd | 1.923 (0.2349) | 1.940 (0.2328)
  12 cpd | 1.527 (0.2793) | 1.558 (0.2566)
  18 cpd | 0.993 (0.2874) | 1.090 (0.2661)

5. Primary Outcome: Mean Photopic With Glare Binocular Distance Contrast Sensitivity
Description: Contrast sensitivity was assessed binocularly with the subject's best spectacle correction under photopic conditions at a distance of 8 feet from the eye at spatial frequencies of 3, 6, and 12, and 18 cpd using the Vector Vision CSV 1000-HGT with a glare source. Raw scores from contrast sensitivity testing were transformed to log units. Subjects who were unable to see a targeted spatial frequency at any available contrast, including that of the reference patch, were assigned the lowest measurable value. A higher numeric value represents better contrast sensitivity. Hypothesis testing was not planned for this outcome measure.
Time Frame: Month 6 (Day 120-180), post second eye implantation
Population: Safety Analysis Set with contrast sensitivity test
Measure: Mean (Standard Deviation); unit: log units
Arm/Group | TFNT00 | SN60AT
Number analyzed (Participants) | 127 | 111
log units
  3 cpd | 1.759 (0.1890) | 1.753 (0.1928)
  6 cpd | 1.897 (0.2322) | 1.971 (0.1952)
  12 cpd | 1.566 (0.2728) | 1.593 (0.2659)
  18 cpd | 1.037 (0.2762) | 1.121 (0.2537)

6. Primary Outcome: Mean Mesopic Without Glare Binocular Distance Contrast Sensitivity
Description: Contrast sensitivity was assessed binocularly with the subject's best spectacle correction under mesopic (dimly-lit) conditions at a distance of 8 feet from the eye at spatial frequencies of 1.5, 3, 6, and 12 cpd using the Vector Vision CSV 1000-HGT without a glare source. Raw scores from contrast sensitivity testing were transformed to log units. Subjects who were unable to see a targeted spatial frequency at any available contrast, including that of the reference patch, were assigned the lowest measurable value. A higher numeric value represents better contrast sensitivity. Hypothesis testing was not planned for this outcome measure.
Time Frame: Month 6 (Day 120-180), post second eye implantation
Population: Safety Analysis Set with contrast sensitivity test
Measure: Mean (Standard Deviation); unit: log units
Arm/Group | TFNT00 | SN60AT
Number analyzed (Participants) | 127 | 111
log units
  1.5 cpd | 1.673 (0.2601) | 1.679 (0.2190)
  3 cpd | 1.717 (0.2397) | 1.689 (0.2177)
  6 cpd | 1.715 (0.2875) | 1.777 (0.2871)
  12 cpd | 1.211 (0.4047) | 1.290 (0.4384)

7. Primary Outcome: Mean Mesopic With Glare Binocular Distance Contrast Sensitivity
Description: Contrast sensitivity was assessed binocularly with the subject's best spectacle correction under mesopic conditions at a distance of 8 feet from the eye at spatial frequencies of 1.5, 3, 6, and 12 cpd using the Vector Vision CSV 1000-HGT with a glare source. Raw scores from contrast sensitivity testing were transformed to log units. Subjects who were unable to see a targeted spatial frequency at any available contrast, including that of the reference patch, were assigned the lowest measurable value. A higher numeric value represents better contrast sensitivity. Hypothesis testing was not planned for this outcome measure.
Time Frame: Month 6 (Day 120-180), post second eye implantation
Population: Safety Analysis Set with contrast sensitivity test
Measure: Mean (Standard Deviation); unit: log units
Arm/Group | TFNT00 | SN60AT
Number analyzed (Participants) | 127 | 111
log units
  1.5 cpd | 1.658 (0.2296) | 1.678 (0.2091)
  3 cpd | 1.709 (0.2307) | 1.692 (0.2089)
  6 cpd | 1.691 (0.3238) | 1.786 (0.2775)
  12 cpd | 1.129 (0.4146) | 1.233 (0.4599)

8. Secondary Outcome: Mean Photopic Monocular Distance Corrected Visual Acuity at Intermediate (66 cm)
Description: VA was tested monocularly under photopic conditions using the manifest refraction adjusted for optical infinity and 100% contrast electronic ETDRS charts at a distance of 66 cm m from the eye. Monocular distance corrected visual acuity at intermediate was measured in logMAR, with 0.02 logMAR increment corresponding to a single letter on an ETDRS chart. A lower numeric value represents better visual acuity. This analysis was prespecified for the first operative eye.
Time Frame: Month 6 (Day 120-180), post second eye implantation
Population: All-Implanted Analysis Set with data at visit
Measure: Least Squares Mean (Standard Error); unit: logMAR
Units Other Than Participants: Eyes
Arm/Group | TFNT00 | SN60AT
Number analyzed (Participants) | 127 | 113
Number analyzed (Eyes) | 127 | 113
logMAR | 0.070 (0.0108) | 0.327 (0.0114)
Statistical Analysis 1: Comparison: TFNT00 vs SN60AT; Test type: Superiority; p < 0.001, Mixed Models Analysis; Least Squares Mean Difference = -0.257, 95% CI 2-sided [-0.287 to -0.227], Standard Error of Mean 0.0153

9. Secondary Outcome: Proportion of Subjects Who Respond "Never" to Question 1 of the Intraocular Lens Satisfaction (IOLSAT) Questionnaire
Description: The IOLSAT is a patient-reported outcomes questionnaire. Subjects were asked, "Overall, in the past 7 days, how often did you need to wear eyeglasses to see?" The proportion of subjects who respond "Never" is reported as a percentage calculated as (# of subjects responding "Never") divided by (# of subjects with bilateral implantation and concordant, non-missing data) times 100.
Time Frame: Month 6 (Day 120-180), post second eye implantation
Population: This analysis population includes all subjects with bilateral implantation and concordant, non-missing data.
Measure: Number; unit: percentage of subjects
Arm/Group | TFNT00 | SN60AT
Number analyzed (Participants) | 123 | 110
percentage of subjects | 80.5 | 8.2
Statistical Analysis 1: Comparison: TFNT00 vs SN60AT; Test type: Superiority; Mantel-Haenszel common difference = 71.2, 95% CI 2-sided [61.87 to 80.46]

10. Secondary Outcome: Rate of Severe Visual Disturbances as Reported by the Subject Using the Questionnaire for Visual Disturbances (QUVID)
Description: QUVID is a patient-reported outcomes questionnaire that collects responses about visual disturbance. Subjects were asked if they experienced any of the visual disturbances in the past 7 days from when the questionnaire was conducted and to answer about how severe their worst experience was on a scale from 0-4, where 0=none and 4=severe. The percentage of subjects responding "Severe" was calculated as (# of subjects responding "Severe") divided by (# of subjects with bilateral implantation and non-missing data in the specified category) times 100. Hypothesis testing was not planned for this outcome measure.
Time Frame: Month 6 (Day 120-180), post second eye implantation
Population: This analysis population includes all subjects with bilateral implantation and non-missing data.
Measure: Count of Participants; unit: Participants
Arm/Group | TFNT00 | SN60AT
Number analyzed (Participants) | 127 | 111
Participants
  Starbursts: number analyzed (Participants) | 125 | 109
  Starbursts | 20 | 2
  Halos: number analyzed (Participants) | 127 | 110
  Halos | 16 | 1
  Glare: number analyzed (Participants) | 126 | 111
  Glare | 4 | 2
  Hazy vision: number analyzed (Participants) | 125 | 110
  Hazy vision | 0 | 0
  Blurred vision | 0 | 0
  Double vision: number analyzed (Participants) | 125 | 110
  Double vision | 0 | 0
  Dark area | 0 | 0

11. Secondary Outcome: Rate of Most Bothersome Visual Disturbances as Reported by the Subject Using the QUVID
Description: Subjects were asked if they experienced any of the visual disturbances in the past 7 days from when the questionnaire was conducted and to answer how much the disturbance bothered them on a scale from 0-4, where 0=not bothered at all and 4=bothered very much. The percentage of subjects with most bothersome visual disturbances was calculated as (# of subjects responding "Bothered very much") divided by (# of subjects with bilateral implantation and non-missing data in the specified category) times 100. Hypothesis testing was not planned for this outcome measure.
Time Frame: Month 6 (Day 120-180), post second eye implantation
Population: This analysis population includes all subjects with bilateral implantation and non-missing data.
Measure: Count of Participants; unit: Participants
Arm/Group | TFNT00 | SN60AT
Number analyzed (Participants) | 127 | 111
Participants
  Starbursts: number analyzed (Participants) | 125 | 109
  Starbursts | 6 | 1
  Halos: number analyzed (Participants) | 127 | 110
  Halos | 3 | 1
  Glare: number analyzed (Participants) | 126 | 111
  Glare | 2 | 1
  Hazy vision: number analyzed (Participants) | 125 | 110
  Hazy vision | 0 | 1
  Blurred vision | 0 | 2
  Double vision: number analyzed (Participants) | 125 | 110
  Double vision | 0 | 0
  Dark area | 0 | 0

ADVERSE EVENTS:
Time Frame: Implantation through study completion, an average of 7 months
Description: Adverse Events (AE) were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator. This analysis population includes all eyes with attempted (successful or aborted after contact with the eye) IOL implantation (Safety Analysis Set). "At Risk" population for ocular AEs is included with unit of "eyes."
Groups:
- Preoperative: All subjects in the safety analysis set prior to initiation of treatment.
- TFNT00 - 1st Eye: All first study eyes implanted with AcrySof IQ PanOptix Multifocal IOL Model TFNT00.
- TFNT00 - 2nd Eye: All second study eyes implanted with AcrySof IQ PanOptix Multifocal IOL Model TFNT00.
- TFNT00 - Systemic: All subjects implanted with AcrySof IQ PanOptix Multifocal IOL Model TFNT00.
- SN60AT - 1st Eye: All first study eyes implanted with AcrySof Monofocal IOL Model SN60AT.
- SN60AT - 2nd Eye: All second study eyes implanted with AcrySof Monofocal IOL Model SN60AT.
- SN60AT - Systemic: All subjects implanted with AcrySof Monofocal IOL Model SN60AT.
Arm/Group | Preoperative | TFNT00 - 1st Eye | TFNT00 - 2nd Eye | TFNT00 - Systemic | SN60AT - 1st Eye | SN60AT - 2nd Eye | SN60AT - Systemic
All-Cause Mortality (participants affected / at risk) | 0/243 | 0/129 | 0/127 | 0/129 | 0/114 | 0/111 | 0/114
Serious Adverse Events (participants affected / at risk) | 0/243 | 2/129 | 2/127 | 4/129 | 2/114 | 1/111 | 3/114
Other Adverse Events (participants affected / at risk) | 1/243 | 24/129 | 24/127 | 0/129 | 10/114 | 7/111 | 0/114
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Preoperative (N=243) | TFNT00 - 1st Eye (N=129) | TFNT00 - 2nd Eye (N=127) | TFNT00 - Systemic (N=129) | SN60AT - 1st Eye (N=114) | SN60AT - 2nd Eye (N=111) | SN60AT - Systemic (N=114)
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Age-related macular degeneration (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Cystoid macular oedema (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Posterior capsule rupture (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vitreous prolapse (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal wall haematoma (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Device dislocation (Product Issues) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Colectomy (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Intra-ocular injection (Surgical and medical procedures) | 0 | 1 | 2 | 1 | 1 | 1 | 0
Intraocular lens repositioning (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lens extraction (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Vitrectomy (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Retinal tear (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Preoperative (N=243) | TFNT00 - 1st Eye (N=129) | TFNT00 - 2nd Eye (N=127) | TFNT00 - Systemic (N=129) | SN60AT - 1st Eye (N=114) | SN60AT - 2nd Eye (N=111) | SN60AT - Systemic (N=114)
Posterior capsule opacification (Eye disorders) | 0 | 17 | 19 | 0 | 4 | 5 | 0
Intraocular pressure increased (Investigations) | 1 | 7 | 5 | 0 | 6 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (2):
  • Study Protocol (2018-03-28): https://cdn.clinicaltrials.gov/large-docs/08/NCT03280108/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-26): https://cdn.clinicaltrials.gov/large-docs/08/NCT03280108/SAP_001.pdf